CLINICAL TRIAL: NCT05081674
Title: Evaluation of Costs and Outcomes of the Implementation of Treatment Protocol Based on Rational Utilization of Anti-PD1 Agents in Patients With Non-small-cell Lung Cancer in the Brazilian Public Health System
Brief Title: Brazilian Lung Immunotherapy Study
Acronym: BLISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4009-19
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2021-10

CONDITIONS: Lung Neoplasm
Keywords: Non-small cell lung cancer; NSCLC; Lung adenocarcinoma; Squamous cell carcinoma of the lung; Immunotherapy; PD-1; Nivolumab; Pembrolizumab
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — alectinib; pembrolizumab; Nivolumab; Erlotinib Hydrochloride

STUDY DESIGN:
Intervention Model Description: Patients are treated in one of 4 different arms based on biomarker testing. There is no randomization or cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ALK-translocated (Active Comparator): 1. st line Alectinib
  2. nd line Carboplatin pemetrexed
  3. rd line Docetaxel
  Interventions: Drug: Alectinib
- EGFR-mutant (Active Comparator): 1. st line Erlotinib
  2. nd line Carboplatin pemetrexed
  3. rd line Docetaxel
  Interventions: Drug: Erlotinib
- PD-L1 >= 50% (Active Comparator): 1. st line Pembrolizumab
  2. nd line Carboplatin pemetrexed
  3. rd line Docetaxel
  Interventions: Drug: Pembrolizumab
- PD-L1< 50% (Active Comparator): 1. st line Carboplatin pemetrexed
  2. nd line nivolumab
  3. rd line Docetaxel
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Alectinib — 600mg 1OD
  Other Names: Alecensa
  Arms: ALK-translocated
Drug: Pembrolizumab — 200mg every 21 days
  Other Names: Keytruda
  Arms: PD-L1 >= 50%
Drug: Nivolumab — 6mg/kg every 4 weeks
  Other Names: Opdivo
  Arms: PD-L1< 50%
Drug: Erlotinib — 150mg
  Other Names: Tarceva
  Arms: EGFR-mutant

SUMMARY:
Immunotherapy with anti-PD-1/PD-L1 agents either as single agents or combined with chemotherapy is now considered the standard of care for patients with non-small-cell lung cancer. However, it has not been incorporated in the Brazilian Public Health System because of concerns about patient eligibility, safety and costs. It is known that simple biomarkers can be used to select patients for immunotherapy, such as EGRF, ALK and PD-L1 status in the tumors. We created a treatment protocol based on these 3 markers and treated 154 patients with non-small-cell-lung cancer in a Public Hospital in Brazil. The goal of this project is to identify the prevalence of these markers in the Brazilian population (to estimate patient eligibility), outcomes and costs of therapy.

DETAILED DESCRIPTION:
Patients with metastatic non-small-cell lung cancer will undergo tumor testing for EGFR (by PCR), ALK and PD-L1 (by immunohistochemistry) and receive therapy based on these results.

* Patients with ALK-translocated tumors will receive first-line therapy with Alectinib, second-line therapy with carboplatin and pemetrexed and third-line therapy with docetaxel
* Patients with EGFR-mutated tumors will receive first-line therapy with Erlotinib, second-line therapy with carboplatin and pemetrexed and third-line therapy with docetaxel
* Patients with ALK/EGFRwt tumors and PD-L1>=50% will receive first-line pembrolizumab, second-line carboplatin-pemetrexed and third line docetaxel
* Patients with ALK/EGFRwt tumors and PD-L1<50% will receive first-line carboplatin-pemetrexed, second-line nivolumab and third line docetaxel.

Therapy costs will be estimated, including hospital admissions and reported for each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIc or IV Non-small cell lung cancer
* Good performance status (ECOG 0-2)
* Available tissue for tumor markers
* Plan to undergo systemic therapy

Exclusion Criteria:

* Inadequate cardiac, renal, liver of bone-marrow function
* Plan to undergo definitive radiation or curative surgery
* Consent withdraw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Total cost of therapy | Up to 3 years after starting systemic therapy
  Sum of all direct costs involved in patient care, including admissions

SECONDARY OUTCOMES:
Median overall survival | Up to 3 years after starting systemic therapy
  Median survival from first systemic therapy
Prevalence of ALK, EGFR, PD-L1>=50% | Up to 3 years after starting systemic therapy
  Prevalence of the 3 biomarkers in an unselected NSCLC population in Brazil

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Gomes, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Municipal Vila Santa Catarina, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web site of the Brazilian Ministry of Health — https://hospitais.proadi-sus.org.br/